CLINICAL TRIAL: NCT07180407
Title: The Post-ICU Pain Study: a Multicenter, Prospective, Inception Cohort Study
Brief Title: The Post-ICU Pain Study
Acronym: PIP
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PIP-study
Record Dates: First submitted 2025-07-15; First posted 2025-09-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Post Intensive Care Unit Syndrome; Quality of Life; Pain Disorder
Keywords: intensive care units; chronic pain; sleep disorder; anxiety and depression; icu survivors
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders; Sleep Wake Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND: ICU survivors may experience serious psychological, physical and cognitive impairments following ICU admission, collectively termed Post Intensive Care Syndrome (PICS). Persistent pain is an underrecognized component of PICS. Previous research has shown that persistent pain is a profound clinical challenge in ICU survivors, however, research demonstrates conflicting results. Furthermore, no studies have examined the prevalence of persistent pain in ICU survivors in a contemporary Danish ICU setting.

OBJECTIVES: We aim to examine the clinical trajectory, risk factors, and pathophysiology of persistent pain in ICU survivors in Denmark.

DESIGN AND SAMPLE SIZE: The study is designed as a multicenter, prospective, inception cohort study with clinical follow-up. Based on the pre-study sample size calculation, 800 patients will be included. Patients will be contacted by telephone 90 days and 180 days after ICU discharge, and a series of questionnaires regarding pain, sleep quality, affective state and quality of life will be completed. A subgroup of patients will undergo a detailed clinical examination including quantitative sensory testing between 180-365 days after ICU discharge.

POPULATION: Patients will be recruited from 4 Danish ICU departments. Inclusion criteria include adult patients (18 years of age), acute admission to the ICU, and an ICU admission of a minimum of 48 hours.

OUTCOMES: The primary outcome is the prevalence of pain assessed by the Brief Pain Inventory (BPI) at 90 and 180 days after ICU discharge. Secondary outcomes include additional detailed descriptions of pain and daily activity, sleep quality, affective state, quality of life, treatment- and patient-related risk factors, and biomarkers associated with development of persistent pain.

Substudies:

- QST substudy: 80 participants (40 with pain and 40 without pain) recruited from the main cohort will undergo Quantative Somatosensory Testing (QST). The objectives are first, to delineate somatosensory profiles of ICU survivors with and without pain, and second, to examine the presence of neuropathic pain in ICU survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients ≥18 years of age
* Acute admission to the ICU
* ICU length of stay of at least 48 hours

Exclusion Criteria:

* Patients transferred from a non-participating ICU
* Patients with pre-planned admission to the ICU e.g., following elective surgery
* Patients unable to complete questionnaires, including those who are unable to understand or speak Danish, or patients with severe cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pain | 180 day follow-up
  Patients are defined as having pain if they answer "yes" to question number 1 in the Brief Pain Inventory - Short Form

SECONDARY OUTCOMES:
Brief Pain Inventory - Short Form (BPI-SF) | At follow-up at 90 and 180 days
  Additional components of the Brief Pain Invenstory Short Form
Incidence of new-onset persistent pain after ICU discharge | at 90 and 180 days follow-up
  Definition of new-onset persistent pain: Individuals presenting with pain according to Brief Pain Inventory Short Form at 90 AND 180 days follow-up AND not suffering from persistent pain/using pain medication regularly before ICU admission, as reported by the individual.
Quality of life measured by EuroQol-5-domain 5-level (EQ-5D-5L) | at 90 and 180 days
  The EQ-5D-5L comprises 5 components (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression) which can be rated at 5 levels. Furthermore, a Visual Analog Scale (VAS) documents self-rated health
The Single Item Sleep Quality Scale (SQS) | at 90 and 180 days
  The respondent is asked to rate the overall quality of sleep over a 7-day recall period on a VAS. Respondents are instructed to consider the following components before answering the questionnaire: hours of sleep, night wakings, how easily they fall asleep, how often they wake earlier then needed, and how refreshed they feel when waking. Sleep quality is scored as follows: 0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent
Hospital Anxiety and Depression Scale (HADS) | at 90 and 180 days
  It comprises seven questions regarding anxiety and seven questions regarding depressive symptoms. Anxiety and depression are scored separately with recommended cut-off values of 8-10 for possible presence of a mood disorder and >11 for probable presence of a mood disorder
Self-Reported Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) | 90 and 180 days
  Only patients answering "yes" to the Brief Pain Inventory Short Form, question number 1, will be asked to fill out the S-LANSS. The tool was created as a clinical tool to identify pain primarily of neuropathic origin, allowing for the differentiation between neuropathic pain and nociceptive pain. It contains 7 items assessing pain quality, sensory changes and specific symptoms commonly associated with neuropathic pain. A score above 12 suggests neuropathic pain
30-day mortality | 30 days
90-day mortality | 90 days
180 days mortality | 180 days

OTHER OUTCOMES:
The Short Physical Performance Battery (SPPB) | between 180 days followup and 360 days.
  QST SUBSTUDY: This test includes a series of tasks designed to examine physical performance. The SPPB requires limited space and takes about 10 minutes to complete. It contains 3 domains (3 m gait speed, 5 times chair stands, and 3 progressive standing balance tasks). Each component is scored separately, and a total score is calculated. The maximum score is 12 indicating little to no mobility impairment
PainDETECT (PD-Q) | between 180 days followup and 360 days
  QST SUBSTUDY: The questionnaire assesses pain intensity (three questions), pain course patterns, the location of pain and presence of radiating pain (via a body chart), and sensory descriptors of pain (seven questions). Scores of 0-12 indicate neuropathic pain component is unlikely, scores of 12-18 indicates results are ambiguous, however a neuropathic component can pe present, and lastly scores of 19-38 indicates neuropathic pain component is likely
QST outcomes | between 180 days followup and 360 days
  QST SUBSTUDY:
  - simple reaction time (seconds)
QST outcomes | between 180 days followup and 360 days
  QST SUBSTUDY:
  - Thermal thresholds: Thresholds are determined by increasing the thermode temperature from baseline 32°C (ramp rate + 1.0 °C/s) until the subject activates the 'stop' button. WDT is defined as the point at which the patient first perceives a sensation of warmth. HPT is defined as the point at which the thermal sensation first turns into pain. The cut-off temperature is 50°C, avoiding the risk of thermal skin injuries
QST outcomes | between 180 days followup and 360 days
  QST SUBSTUDY:
  - Pinprick thresholds and temporal summation (mN)
QST outcomes | between 180 days followup and 360 days
  QST SUBSTUDY:
  - Offset analgesia (numeric rating scale; 0-100).
QST outcomes | between 180 days followup and 360 days
  QST SUBSTUDY:
  - Conditioned pain modulation (seconds): includes the cold pressor test (CPT; conditioning stimulus) and pressure algometry (test stimulus).

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Zealand University Hospital, Køge
  - Zealand University Hospital, Nykøbing Falster
  - Zealand University Hospital, Roskilde